CLINICAL TRIAL: NCT05535972
Title: A 12-week, Prospective, Open Label, Single Cohort Study to Evaluate the Real-world Effectiveness of Fluticasone Furoate/Umeclidinium Bromide/Vilanterol in a Single Inhaler (Trelegy Ellipta) in Symptomatic Chronic Obstructive Pulmonary Disease (COPD) Patients
Brief Title: To Evaluate Real-World Effectiveness of Fluticasone Furoate/Umeclidinium Bromide/Vilanterol (FF/UMEC/VI) in a Single Inhaler (Trelegy Ellipta) in Participants With Symptomatic COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 217658
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: TRELEGY ELLIPTA; Single Inhaler; Fluticasone Furoate; Umeclidinium Bromide; Vilanterol; FF/UMEC/VI
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants receiving TRELEGY ELLIPTA (Experimental): Participants will receive FF/UMEC/VI, inhalation powder, once daily, in a single device (TRELEGY ELLIPTA) for 12 weeks.
  Interventions: Drug: FF/UMEC/VI

INTERVENTIONS:
Drug: FF/UMEC/VI — FF/UMEC/VI will be administered in a single inhaler Trelegy Ellipta.
  Other Names: TRELEGY ELLIPTA

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of TRELEGY ELLIPTA on health status in participants with symptomatic COPD. The secondary objective is to evaluate the effectiveness of TRELEGY ELLIPTA on dyspnea and lung function in participants with symptomatic COPD. TRELEGY and ELLIPTA are trademarks of the GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 40 years or above of age inclusive, at the time of signing the informed consent.
* Participants with a documented physician diagnosis of COPD.
* CAT greater than or equal to (≥) 10.
* Existing COPD Maintenance Treatment. Participants currently receiving one of the maintenance therapies given below who have been prescribed it continually for at least 12 weeks prior to screening (Visit 1): Inhaled Corticosteroids/ Long-Acting Beta-2-Agonists (ICS/LABA) (single or multiple inhalers); Long-Acting Muscarinic Antagonist (LAMA)/LABA (single or multiple inhalers); Free combination of inhaled corticosteroids (ICS), LAMA, LABA.
* Current or former cigarette smokers with a history of cigarette smoking history ≥10 pack-years at screening.
* Trelegy is prescribed under the discretion of clinical physicians with medical records providing documentation of a Trelegy prescription in daily practice.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Prescribed with Trelegy within one year prior to screening (Visit 1).
* Participants who, in the opinion of the treating investigator, are chronic users of oral corticosteroids for respiratory or other indications (if unsure discuss with the medical monitor prior to screening). Chronic use is defined as more than 14 days continuous use during the 12 weeks prior to Visit 1.
* Participants with any life-threatening condition i.e. low probability, in the opinion of the investigator, of 3-month survival due to severity of COPD or comorbid condition.
* Participants with unstable COPD. Participants with resolution of an exacerbation less than 2 weeks prior to Visit 1. Participants may be rescreened 2 weeks after resolution of exacerbation (exacerbation is defined as: requiring treatment with antibiotics and/or systemic steroids or hospitalization; resolution is defined as: 2 weeks after all symptoms have resolved and any medicines to treat the exacerbation have finished).
* Participants who need more than 3 liter per minute (L/min) supplemental oxygen at rest at screening.
* Other diseases/abnormalities: Participants with historical or current evidence of uncontrolled or clinically significant disease. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the participant at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Participant received any investigational drug in other clinical trial within four weeks or 5 half-lives prior to this study whichever is longer.
* Any conditions or illnesses listed in the section of contraindications in the Summary of Product Characteristics (SmPC) of Trelegy, i.e., hypersensitivity to the active substances of TRELEGY ELLIPTA.
* Participants with known COVID-19 positive contacts within the past 14 days.
* Inability to read: In the opinion of the Investigator, any participant who is unable to read and/or would not be able to complete study related materials.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Dongguan, China

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Ma J, Dou F, Zhou W, Li L, Zhu J, Zhang Y, Zhou L, Su L, Dong L, He Y, Ye A, Slade D, Zheng J. Real-world effectiveness of single-inhaler fluticasone furoate/umeclidinium bromide/vilanterol in Chinese patients with symptomatic chronic obstructive pulmonary disease (COPD): a post-marketing, prospective, multicenter, observational study. Curr Med Res Opin. 2025 Jul;41(7):1363-1372. doi: 10.1080/03007995.2025.2536600. Epub 2025 Jul 29. PMID 40704458

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 463 participants were enrolled in this study, however only 460 participants (3 participants were never dosed) were dosed into the study to receive Trelegy creating the Full Analysis Set (FAS) (All participants who were enrolled into the study and took at least one dose of Trelegy).
Groups:
- Trelegy (FF/UMEC/VI ELLIPTA): Participants with symptomatic chronic obstructive pulmonary disease (COPD) received a single dose of Trelegy (fluticasone furoate [FF] 100 microgram [ug] / umeclidinium [UMEC] 62.5 ug / vilanterol [VI] 25 ug) in a single inhaler (TRELEGY ELLIPTA) via inhalation for 12 weeks.
Period: Overall Study
Arm/Group | Trelegy (FF/UMEC/VI ELLIPTA)
Started (Enrolled) | 463
Full Analysis Set | 460
Completed | 419
Not Completed | 44
Not completed — Withdrawal by Subject | 31
Not completed — Lost to Follow-up | 5
Not completed — Adverse Event | 6
Not completed — Protocol Deviation | 2

BASELINE CHARACTERISTICS:
Population: Baseline Characteristic data are reported for the Full Analysis Set (FAS) which included all participants who were enrolled into the study and took at least one dose of Trelegy.
Arm/Group | Trelegy (FF/UMEC/VI ELLIPTA)
Number analyzed (Participants) | 460
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.74 (8.118)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 434
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 460
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in COPD Assessment Test (CAT) Score at Week 12
Description: The CAT is a validated 8-items questionnaire developed for use in routine clinical practice to measure the health status of participants with COPD. Participants rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment), higher score indicates greater impairment. A total CAT score was calculated by summing the non-missing scores of the eight items with a scoring range of 0 (no disease impact) to 40 (maximum disease impact). Higher scores indicated greater disease impact. Baseline was defined as the latest pre-dose of Trelegy assessment with a non-missing value, including those from unscheduled visits. Change from Baseline (CFB) was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, pre-dose) and at Week 12
Population: Full Analysis Set included all participants who were enrolled into the study and took at least one dose of Trelegy. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the 'Overall Number of Participants Analyzed' field.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Trelegy (FF/UMEC/VI ELLIPTA)
Number analyzed (Participants) | 422
Scores on a scale | -6.8 (5.49)
Statistical Analysis 1: Comparison: Trelegy (FF/UMEC/VI ELLIPTA); Test type: Other; Least Square Mean = -6.81, 95% CI 2-sided [-7.28 to -6.33], Standard Error of Mean 0.241 — CFB in CAT score was analyzed using Mixed Model Repeated Measures(MMRM) model with covariates of smoking status, CAT score at Baseline, visit, interaction of CAT score at Baseline*visit. Estimates derived from inverse probability weighted MMRM model

2. Secondary Outcome: Change From Baseline in Modified Medical Research Council (mMRC) Grading System at Week 12 (Patient Version)
Description: mMRC(Patient Version[Pt.V]) was used to assess breathlessness state of participant before and after treatment. mMRC (Pt V) was completed by each participant firstly, without supervision.Participants were scored on a scale of 0 (no impact) to 4(worst possible impact) depending on their disability due to shortness of breath. Higher scores indicated greater disease impact;where 0=only get breathless with strenuous exercise;1=get short of breath when hurrying on the level/walking up a slight hill;2=walk slower than people of same age on the level because of breathlessness/have to stop for breath when walking at own pace on the level;3=stop for breath after walking about 100 yards/after a few minutes on the level;4=too breathless to leave house/breathless when dressing. Baseline=latest pre-dose of Trelegy assessment with a non-missing value, including those from unscheduled visits. Change from Baseline=post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, pre-dose) and at Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Trelegy (FF/UMEC/VI ELLIPTA)
Number analyzed (Participants) | 422
Scores on a scale | -0.5 (0.91)

3. Secondary Outcome: Change From Baseline in Modified Medical Research Council (mMRC) Dyspnea Scale at Week 12 (Physician Version)
Description: mMRC(Physician Version[PV]) was used to assess breathlessness state of participant before and after treatment. Physicians completed mMRC(PV) through their observation. Participants were scored on a scale of 0 (no impact) to 4(worst possible impact) depending on their disability due to shortness of breath. Higher scores indicated greater disease impact; where 0=no breathlessness except on strenuous exercise; 1=shortness of breath when hurrying on the level ground or walking up a slight hill; 2=walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3=stops for breath after walking about 100 yards or after few minutes on level ground; 4=too breathless to leave house or breathless when dressing or undressing. Baseline=latest pre-dose of Trelegy assessment with a non-missing value, including those from unscheduled visits. Change from Baseline=post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, pre-dose) and at Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Trelegy (FF/UMEC/VI ELLIPTA)
Number analyzed (Participants) | 422
Scores on a scale | -0.5 (0.89)

4. Secondary Outcome: Change From Baseline in Pre-dose Forced Expiratory Volume in 1 Second (FEV1) at Week 12
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. FEV1 was measured using spirometry. Baseline was defined as the latest pre-dose of Trelegy assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, pre-dose) and at Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Trelegy (FF/UMEC/VI ELLIPTA)
Number analyzed (Participants) | 411
Liters | 0.132 (0.2897)

5. Secondary Outcome: Percentage of Participants Having >=2 Unit Decrease in CAT Score From Baseline at Week 12
Description: The CAT is a validated 8-items questionnaire developed for use in routine clinical practice to measure the health status of participants with COPD. Participants rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment), higher score indicates greater impairment. A total CAT score was calculated by summing the non-missing scores of the eight items with a scoring range of 0 (no disease impact) to 40 (maximum disease impact). Higher scores indicated greater disease impact. Baseline was defined as the latest pre-dose of Trelegy assessment with a non-missing value, including those from unscheduled visits. Percentage values are rounded-off. Percentage of participants having >=2 unit decrease in CAT score from Baseline at week 12 has been presented.
Time Frame: Baseline (Day 1, pre-dose) and at Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trelegy (FF/UMEC/VI ELLIPTA)
Number analyzed (Participants) | 422
Percentage of Participants | 86.0 [82.7 to 89.3]

6. Secondary Outcome: Change From Baseline in COPD Assessment Test (CAT) Score at Week 4
Description: as for outcome 1
Time Frame: Baseline (Day 1, pre-dose) and at Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Trelegy (FF/UMEC/VI ELLIPTA)
Number analyzed (Participants) | 439
Scores on a scale | -4.4 (5.29)

7. Secondary Outcome: Number of Participants With Trelegy Related Non-serious Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 251 days
Population: Full Analysis Set included all participants who were enrolled into the study and took at least one dose of Trelegy.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelegy (FF/UMEC/VI ELLIPTA)
Number analyzed (Participants) | 460
Participants | 9

8. Secondary Outcome: Number of Participants With Trelegy Related Serious Adverse Events (SAEs)
Description: A SAE is defined as any serious adverse event that, at any dose; results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, a suspected transmission of any infectious agent via an authorized medicinal product or other situations as judged by physician.
Time Frame: Up to 251 days
Population: Full Analysis Set included all participants who were enrolled into the study and took at least one dose of Trelegy.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelegy (FF/UMEC/VI ELLIPTA)
Number analyzed (Participants) | 460
Participants | 1

9. Secondary Outcome: Number of Participants With Trelegy Related AEs Leading to the Discontinuation
Description: as for outcome 7
Time Frame: Up to 251 days
Population: Full Analysis Set included all participants who were enrolled into the study and took at least one dose of Trelegy.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelegy (FF/UMEC/VI ELLIPTA)
Number analyzed (Participants) | 460
Participants | 5

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (non-SAEs) and serious adverse events (SAEs) were collected up to 251 days
Description: All-cause mortality, serious adverse events and non-serious adverse events were reported for the Full Analysis Set (FAS). FAS included all participants who were enrolled in the study and took at least one dose of Trelegy. Three participants from Enrolled Population (N=463) did not receive study treatment, hence was not included in FAS Population (N=460).
Arm/Group | Trelegy (FF/UMEC/VI ELLIPTA)
All-Cause Mortality (participants affected / at risk) | 2/460
Serious Adverse Events (participants affected / at risk) | 19/460
Other Adverse Events (participants affected / at risk) | 10/460
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trelegy (FF/UMEC/VI ELLIPTA) (N=460)
COVID-19 (Infections and infestations) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Cerebral thrombosis (Nervous system disorders) | 1 (1)
Intracranial mass (Nervous system disorders) | 1 (1)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trelegy (FF/UMEC/VI ELLIPTA) (N=460)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT05535972/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT05535972/SAP_001.pdf